CLINICAL TRIAL: NCT04581200
Title: Addressing Psychological Distress Symptoms Among Serious Illness Survivors of a Viral Pandemic With a Completely Self-directed, Symptom-responsive Mobile Mindfulness Intervention: a Randomized Controlled Trial
Brief Title: Lift Mobile Mindfulness for COVID-19 Distress Symptoms
Acronym: LIFTCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00106306; 3U01AT009974-03S1 (NIH)
Record Dates: First submitted 2020-10-04; First posted 2020-10-09 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: COVID-19; Cardiorespiratory Failure
Keywords: critical illness; psychological distress; depression; anxiety; adults
MeSH Terms: conditions — COVID-19; Critical Illness; Depression; Anxiety Disorders | interventions — Lifting

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to group assignment, as will the investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lift mobile mindfulness program (Experimental): Will receive standard dose Lift mobile mindfulness program intervention content, app-based response to elevated symptoms, and no introductory call from a therapist. This program lasts 1 month and includes 4 unique weeks' worth of audio, video, and text content.
  Interventions: Behavioral: Lift
- Usual care control (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Lift — The intervention is a mobile app-based mindfulness training program designed to be used over a 1-month period.
  Arms: Lift mobile mindfulness program

SUMMARY:
This is a randomized clinical trial (RCT) nested within the NIH PETAL Network's COVID cohort study (BLUE CORAL [Biology and Longitudinal Epidemiology: COVID Observational Study]) of patients hospitalized for COVID-19-related illness. COVID-19 patients enrolled in BLUE CORAL with elevated distress symptoms 1 month post-discharge will be randomized to either the Lift mobile app intervention or a usual care control.

DETAILED DESCRIPTION:
The novel coronavirus (COVID-19) pandemic has changed access to and the delivery of medical care across the world rapidly and radically as increasingly large waves of patients fill clinics, hospital wards, and intensive care units (ICUs). Patients with comparable illnesses have high rates of persistent psychological distress symptoms including depression, anxiety, and PTSD. Currently there are few easily accessible therapies available for this distress in this time of deep fear and worry, social distancing, cancelled clinics, isolation and quarantine practices, and understaffed hospitals.

Lift, a novel mobile app-based mindfulness intervention, may be able to address COVID-19 patients' distress and access to care issues. Lift was piloted successfully in the intensive care unit (ICU; R34 AT00819) and is currently in the midst of a multicenter factorial experimental clinical trial designed to determine which of 8 versions is optimized for symptom relief, cost, and scalability (parent U01 AT009974).

This 2-arm, parallel group randomized clinical trial seeks to expand the scope of the parent U01 project to test the clinical impact of a psychological distress intervention rapidly deployed during a pandemic. This trial will include 300 patients who were hospitalized due to COVID-19; collect data at 1, 3, and 6 months post-discharge; and address 3 specific aims: (1) Compare the clinical impact of Lift vs. usual care control and (2) Compare long-term (6-month) outcomes of RCT patients both by treatment arm as well to the entire BLUE CORAL cohort, and (3) Explore participant-reported barriers and facilitators to intervention deployment, uptake, and engagement in a pandemic.

ELIGIBILITY:
BLUE CORAL eligibility (the parent cohort study from which RCT participants will be recruited)

Inclusion criteria:

1. Adult hospitalized within 14 days of a positive PCR test for COVID-19
2. Evidence of acute COVID-19, with fever or respiratory manifestations, as characterized by signs and symptoms such as cough, dyspnea, tachypnea, hypoxemia, and infiltrates on chest imaging.

Exclusion criteria:

1. Lack of informed consent
2. More than 72 hours of continuous hospitalization.
3. Comfort care orders in place at the time of enrollment and/or unexpected to survive for 24 hours
4. Prisoners
5. Previous enrollment in BLUE CORAL

LIFT COVID RCT eligibility

Inclusion criteria:

1. Enrolled in BLUE CORAL
2. Survival to time of BLUE CORAL 1-month post-discharge interview

2. English-speaking 3. Domiciled with access to a working telephone and smartphone, tablet, or computer with wifi or internet connection 4. Absence of severe dementia or cognitive dysfunction either before hospitalization or at time of 1 month post-discharge interview

Exclusion criteria:

1. PHQ-9 <5 at time of interview 1 month post-discharge
2. Suicidal ideation at time of interview 1 month post-discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Cox, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - University of Colorado - Denver, Aurora, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Sciences University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
We will follow NIH/NCCIH guidelines for data access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We will follow NIH guidelines.
Access Criteria: We will follow NIH and institutional guidelines.

REFERENCES:
- [Background] Cox CE, Porter LS, Buck PJ, Hoffa M, Jones D, Walton B, Hough CL, Greeson JM. Development and preliminary evaluation of a telephone-based mindfulness training intervention for survivors of critical illness. Ann Am Thorac Soc. 2014 Feb;11(2):173-81. doi: 10.1513/AnnalsATS.201308-283OC. PMID 24303911
- [Background] Cox CE, Hough CL, Jones DM, Ungar A, Reagan W, Key MD, Gremore T, Olsen MK, Sanders L, Greeson JM, Porter LS. Effects of mindfulness training programmes delivered by a self-directed mobile app and by telephone compared with an education programme for survivors of critical illness: a pilot randomised clinical trial. Thorax. 2019 Jan;74(1):33-42. doi: 10.1136/thoraxjnl-2017-211264. Epub 2018 May 23. PMID 29793970
- [Background] Cox CE, Olsen MK, Gallis JA, Porter LS, Greeson JM, Gremore T, Frear A, Ungar A, McKeehan J, McDowell B, McDaniel H, Moss M, Hough CL. Optimizing a self-directed mobile mindfulness intervention for improving cardiorespiratory failure survivors' psychological distress (LIFT2): Design and rationale of a randomized factorial experimental clinical trial. Contemp Clin Trials. 2020 Sep;96:106119. doi: 10.1016/j.cct.2020.106119. Epub 2020 Aug 15. PMID 32805434
- [Derived] Cox CE, Gallis JA, Olsen MK, Porter LS, Gremore TM, Iwashyna TJ, Caldwell ES, Greeson JM, Moss M, Hough CL. Mobile App-Based Mindfulness Intervention for Addressing Psychological Distress Among Survivors of Hospitalization for COVID-19 Infection. CHEST Crit Care. 2024 Jun;2(2):100063. doi: 10.1016/j.chstcc.2024.100063. Epub 2024 Mar 4. PMID 38957856
- See also: Study website — http://lift.duke.edu/covid

RESULTS

PARTICIPANT FLOW:
Groups:
- Lift Mobile Mindfulness Program: Will receive standard Lift mobile mindfulness program intervention content, app-based response to elevated symptoms, and no introductory call from a therapist. This program lasts 1 month and includes 4 unique weeks' worth of audio, video, and text content.
  Lift: The intervention is a mobile app-based mindfulness training program designed to be used over a 1-month period.
Period: Overall Study
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Started | 29 | 27
Completed | 23 | 22
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (14.2) | 53.1 (11.8) | 51.0 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 19 | 23 | 42
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 14 | 17 | 31
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Health Questionnaire-9 Item Scale (PHQ-9) Over 3 Months Post-discharge
Description: Depression symptoms. Scores range from 0 (better) to 27 (worse)
Time Frame: T1 (time of randomization [i.e., 1 month post-hospital discharge), T2 (2 months post-randomization [i.e., 3 months post-hospital discharge)
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale | 0.09 (3.22) | -0.50 (4.31)
Statistical Analysis 1: Comparison: Lift Mobile Mindfulness Program vs Usual Care Control; Test type: Superiority; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-1.63 to 2.80]

2. Secondary Outcome: Change in Patient Health Questionnaire-9 Item Scale (PHQ-9) Over 6 Months Post-discharge
Description: Depression symptoms. Scores range from 0 (better) to 27 (worse)
Time Frame: T1 (time of randomization [i.e., 1 month post-hospital discharge), T3 (5 months post-randomization [i.e., 6 months post-hospital discharge)
Population: Data not collected on 4 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Number analyzed (Participants) | 27 | 25
score on a scale | -0.63 (5.76) | -0.84 (4.71)
Statistical Analysis 1: Comparison: Lift Mobile Mindfulness Program vs Usual Care Control; Test type: Other — This is an exploratory pilot trial; p = 0.89, t-test, 2 sided; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-2.66 to 3.08]

3. Secondary Outcome: Change in Generalized Anxiety Disorder 7-item Scale (GAD-7) at 3 Months Post-discharge
Description: Anxiety symptoms. Scores range from 0 (better) to 21 (worse).
Time Frame: as for outcome 1
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale | 0.09 (4.76) | -0.27 (5.29)
Statistical Analysis 1: Comparison: Lift Mobile Mindfulness Program vs Usual Care Control; Test type: Superiority; p = 0.81, t-test, 2 sided; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [-2.58 to 3.30]

4. Secondary Outcome: Change in Generalized Anxiety Disorder 7-item Scale (GAD-7) at 6 Months Post-discharge
Description: Anxiety symptoms. Scores range from 0 (better) to 21 (worse).
Time Frame: as for outcome 2
Population: Data not collected on 4 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Number analyzed (Participants) | 27 | 25
score on a scale | 0.26 (4.83) | 0.68 (4.57)
Statistical Analysis 1: Comparison: Lift Mobile Mindfulness Program vs Usual Care Control; Test type: Superiority; p = 0.75, t-test, 2 sided; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-2.98 to 2.14]

5. Secondary Outcome: Change in EuroQOL-5DL (Quality of Life) Scale at 3 Months Post-discharge
Description: EuroQOL-5DL health states can be represented by a single summary number (index value), which reflects how good or bad a health state is according to the preferences of the general population of a country/region. An EQ-5D summary index is derived by applying a formula that attaches values (weights) to each of the levels in each dimension. The index is calculated by deducting the appropriate weights from 1, the value for full health. A higher index value indicates a greater health state; an increase in index value indicates an improvement in health state. The summary item can range from 0 (worst quality of life) to 100 (best quality of life).
Time Frame: as for outcome 1
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: index value
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Number analyzed (Participants) | 23 | 22
index value | 0.02 (0.19) | -0.03 (0.25)
Statistical Analysis 1: Comparison: Lift Mobile Mindfulness Program vs Usual Care Control; Test type: Superiority; p = 0.45, t-test, 2 sided; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.57 to 0.74]

6. Secondary Outcome: Change in EuroQOL-5DL (Quality of Life) Scale at 6 Months Post-discharge
Description: as for outcome 5
Time Frame: as for outcome 2
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: index value
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Number analyzed (Participants) | 23 | 22
index value | 0.6 (0.36) | 0.66 (0.28)
Statistical Analysis 1: Comparison: Lift Mobile Mindfulness Program vs Usual Care Control; Test type: Superiority; p = 0.98, t-test, 2 sided; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-0.13 to 0.13]

7. Secondary Outcome: Number of Participants With Cardiopulmonary Symptoms at 3 Months Post-discharge
Description: Cardiopulmonary symptoms such as breathlessness, fatigue, oxygen use
Time Frame: as for outcome 1
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Number analyzed (Participants) | 23 | 22
Participants | 10 | 4
Statistical Analysis 1: Comparison: Lift Mobile Mindfulness Program vs Usual Care Control; Test type: Superiority; p = 0.08, Fisher Exact

8. Secondary Outcome: Number of Participants With Cardiopulmonary Symptoms at 6 Months Post-discharge
Description: Cardiopulmonary symptoms such as breathlessness, fatigue, oxygen use
Time Frame: as for outcome 2
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Number analyzed (Participants) | 23 | 22
Participants | 8 | 9
Statistical Analysis 1: Comparison: Lift Mobile Mindfulness Program vs Usual Care Control; Test type: Superiority; p = 0.69, Fisher Exact

9. Other Pre Specified Outcome: Healthcare Utilization
Description: Hospital readmissions and clinic visits during follow up
Time Frame: T1 (time of randomization [i.e., 1 month post-hospital discharge), T2 (2 months post-randomization [i.e., 3 months post-hospital discharge), T3 (5 months post-randomization [i.e., 6 months post-hospital discharge)
Population: Data not collected.
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Intervention Adherence as Measured by Percentage of Tasks Completed
Description: Tasks include intervention sessions, weekly surveys, and intervention elements (e.g., videos, audio).
Time Frame: T3 (5 months post-randomization [i.e., 6 months post-hospital discharge)
Population: Not applicable to the usual care arm.
Measure: Mean (Standard Deviation); unit: percentage of tasks completed
Arm/Group | Lift Mobile Mindfulness Program
Number analyzed (Participants) | 23
percentage of tasks completed | 23.0 (29.3)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Hospitalization
Arm/Group | Lift Mobile Mindfulness Program | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT04581200/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT04581200/ICF_000.pdf